CLINICAL TRIAL: NCT01273883
Title: A Phase III Trial of Magnesium Dependent Tinnitus
Brief Title: A Trial of Magnesium Dependent Tinnitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Cevette, Associate Professor of Audiology, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 09-008292
Record Dates: First submitted 2011-01-07; First posted 2011-01-11 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Tinnitus
Keywords: hearing; magnesium
MeSH Terms: conditions — Tinnitus | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium first, then placebo (Experimental): Magnesium 532 mg daily for 25 days followed by 2 weeks of washout followed by 25 days of placebo.
  Interventions: Dietary Supplement: Magnesium; Other: Placebo
- Placebo first, then magnesium (Placebo Comparator): Placebo daily for 25 days followed by 2 weeks of washout followed by magnesium 532 mg daily for 25 days.
  Interventions: Dietary Supplement: Magnesium; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium — Magnesium 532 mg a day
Other: Placebo — matching form/dosage

SUMMARY:
The purpose of this study was to examine any potential benefit in lessening the severity of tinnitus (ringing or booming sensation in one or both ears) in subjects supplemented with magnesium (532 mg daily).

DETAILED DESCRIPTION:
Descriptions of tinnitus date back to the time of ancient Egypt, yet science has failed to unravel the mysterious underlying mechanisms that produce these subjective auditory perceptions of sound. These perceptions may be manifestations of damage resulting from noise exposure, ototoxicity, or other abnormal conditions of the auditory system. However, many individuals have idiopathic tinnitus for which no specific cause can be determined. Although often presenting in conjunction with hearing loss, the magnitude of hearing loss does not necessarily correspond with the severity of tinnitus. In addition, some individuals reporting tinnitus experience concomitant hyperacusis. This relationship suggests these processes may be linked by underlying imbalances at the level of the hair cell. The possible influence of magnesium (Mg) and its antagonist, calcium, has been discussed in the literature as a contributing factor in the mitigation of noise-induced hearing loss, ototoxicity, and the hyperexcitability of the auditory system. Permanent and temporary changes in auditory function have been linked to nutritional deficiencies of magnesium. Mg deficiency has resulted in increased susceptibility to noise-induced hearing loss, ototoxicity, and hyperexcitability of the auditory system.

The recommended daily allowance (RDA) for Mg in adults is 4.5 mg/kg; however, all age groups of Americans fall short of the RDA for Mg by 100 mg daily. This lack of appropriate magnesium intake may have negative consequences. For example, the putative Mg mechanism within the auditory system involves a metabolic cellular cascade of events. Specifically, Mg deficiency leads to increased permeability of the calcium channel in the hair cells with a consequent over-influx of calcium, an increased release of glutamate via exocytosis, and overstimulation of N-methyl-D-aspartate receptors on the auditory nerve fibers. Recent studies of both noise-induced hearing loss and idiopathic sensorineural hearing loss have suggested that Mg supplementation may lessen the severity of tinnitus in patients. Mg improved hearing recovery and lessened tinnitus in patients with idiopathic sudden hearing loss. More recently, a well-controlled study that Mg was a relatively safe and convenient adjunct to corticosteroid treatment for enhancing the improvements of hearing in acute-onset sensorineural hearing loss at a dose of 4 g. The protective effect of Mg in noise-induced hearing loss has been previously reported.

Despite these encouraging findings, no controlled study has examined the effect of Mg supplementation for subjects with moderate to severe tinnitus.

In this study subjects made 4 visits to the clinic over about 2 months. At the first visit, subjects had a hearing test. Prior to beginning each round of supplements, subjects were asked to rate the severity of their tinnitus on a 1-10 scale, and to complete the Tinnitus Handicap Inventory (THI) questionnaire. Subjects were then randomized to 1 of 2 groups. One group began with 532 mg of Mg for 25 days, the other group began with a placebo supplement for 25 days.

At visit 2, the subjects had a hearing test, rated their tinnitus, and completed the THI questionnaire as well as the Treatment Period Survey. Subjects did not take any supplement for 2 weeks, then returned for visit 3.

At Visit 3, the subjects had a hearing test, rated their tinnitus, and completed the THI questionnaire they then took the opposite supplement (placebo or Mg) for 25 days.

At Visit 4, the subjects had a hearing test, rated their tinnitus, and completed the THI questionnaire as well as the Treatment Period Survey.

ELIGIBILITY:
Inclusion criteria:

* Normal Kidney function (last checked within 6 months). Serum creatinine levels 1.5 mg/dL or below for females, 2.0 mg/dL for males.
* An audiogram within the past 6 months
* Mayo Clinic patients who live in Phoenix area

Exclusion criteria:

* Any participant with decreased kidney function within past 6 months, over 1.5 mg/dL for females and over 2.0 mg/dL for males.
* Current treatment with Lithium
* Tinnitus rating with 0, 1, or 2 on the 0-10 Tinnitus scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cevette, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Background] Cevette MJ, Barrs DM, Patel A, Conroy KP, Sydlowski S, Noble BN, Nelson GA, Stepanek J. Phase 2 study examining magnesium-dependent tinnitus. Int Tinnitus J. 2011;16(2):168-73. PMID 22249877

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Magnesium First, Then Placebo | Placebo First, Then Magnesium
Started | 19 (Received at least 1 dose of study drug.) | 19 (Received at least 1 dose of study drug.)
Completed | 17 | 18
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1
Period: Washout Period of 2 Weeks
Arm/Group | Magnesium First, Then Placebo | Placebo First, Then Magnesium
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Magnesium First, Then Placebo | Placebo First, Then Magnesium
Started | 17 | 18
Completed | 15 | 17
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive magnesium first and placebo first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.45 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Distress Rating
Description: This is a single-item patient-reported distress rating on a 0-10 scale, with 0=no tinnitus to 10=worst possible tinnitus.
Time Frame: Pre-treatment, Post-treatment, up to four weeks
Population: Not all subjects completed the distress rating scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Magnesium: Magnesium 532 mg administered daily in either first intervention period or second intervention period.
- Placebo: Placebo administered daily in either first intervention period or second intervention period.
Arm/Group | Magnesium | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale
  Pre-treatment | 5.71 (1.94) | 5.82 (1.94)
  Post-treatment | 5.36 (2.30) | 5.46 (1.99)

2. Secondary Outcome: Comparison of Average Tinnitus Handicap Inventory (THI) Across All Subjects
Description: The Tinnitus Handicap Inventory measures the extent that tinnitus interferes with daily activities and sleep.The questionnaire consists of 25 questions, the score can range from 0 (slight problem) to 100 (catastrophic). The score can be converted to a categorical variable as follows: 0-16=Slight; 18-36=Mild; 38-56=Moderate; 58-76=Severe; 78-100=Catastrophic.
Time Frame: Pre-treatment, Post-treatment, up to four weeks
Population: Not all subjects completed the THI questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Magnesium | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale
  Pre-treatment | 25.7 (22.2) | 25.7 (19.4)
  Post-treatment | 24.1 (19.9) | 23.2 (17.4)

3. Secondary Outcome: Comparison of Average Tinnitus Handicap Inventory (THI) Across All Men
Description: as for outcome 2
Time Frame: Pre-treatment, Post-treatment, up to four weeks
Population: Not all male subjects completed the THI questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Magnesium | Placebo
Number analyzed (Participants) | 19 | 19
units on a scale
  Pre-treatment | 29.1 (24.7) | 27.2 (22.0)
  Post-treatment | 27.8 (21.5) | 25.3 (19.6)

4. Secondary Outcome: Comparison of Average Tinnitus Handicap Inventory (THI) Across All Women
Description: as for outcome 2
Time Frame: Pre-treatment, Post-treatment, up to four weeks
Population: Not all the female subjects completed the THI questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Magnesium | Placebo
Number analyzed (Participants) | 9 | 9
units on a scale
  Pre-treatment | 18.7 (14.7) | 22.6 (12.7)
  Post-treatment | 16.4 (14.4) | 18.4 (10.9)

ADVERSE EVENTS:
Time Frame: Tinnitus patients who presented to the Ear, Nose, and Throat (ENT) department of the Mayo Clinic in Arizona from 2009 to 2012 were screened and asked to participate.
Description: Adverse events during the study will be reported to the study team by the research coordinator who will query the subjects as part of each study visit.
Arm/Group | Magnesium | Placebo
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 7/38 | 3/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium (N=38) | Placebo (N=38)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Elevated Blood Pressure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Loose Stool (Gastrointestinal disorders) | 3 (3) | 1 (1)
Lower Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Emergency Room Visit (General disorders) | 1 (1) | 1 (1)
Intermittent Ankle Swelling (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes